CLINICAL TRIAL: NCT06143605
Title: Clinical Relevance of the Salvage Treatment for Colorectal Neuroendocrine Tumors Based on the Pathological Evaluation Following Initial Endoscopic Resection: A Multi-center Study
Brief Title: Clinical Relevance of the Salvage Treatment for Colorectal Neuroendocrine Tumors
Status: Completed | Type: Observational
Sponsor: Yanhong Deng (Other)
Responsible Party: Sponsor-Investigator, Yanhong Deng, M.D., Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Other Study IDs: GIH-SYip33
Record Dates: First submitted 2023-11-16; First posted 2023-11-22 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Rectal Neoplasms; Neuroendocrine Tumors
Keywords: endoscopic resection
MeSH Terms: conditions — Rectal Neoplasms; Neuroendocrine Tumors | interventions — Salvage Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- salvage treatment group: patients with salvage treatment after endoscopic resection were diagnosed as having positive resection margin status
  Interventions: Procedure: salvage treatment
- without salvage treatment group: patients without salvage treatment after endoscopic resection were diagnosed as having positive resection margin status

INTERVENTIONS:
Procedure: salvage treatment — salvage radical surgery or endoscopic resection
  Groups: salvage treatment group

SUMMARY:
we evaluated all related clinical and pathologic data of rectal NET cases, including the resection margin status, NET grading, and lymphovascular invasion status. Finally, the present study was aimed at (1) determining the risk factors for LN and distant metastases in colorectal NETs (2) clarifying the clinical significance of the salvage treatment for colorectal neuroendocrine tumors following initial endoscopic resection with positive resection margin status and (3) compare different salvage treatment of this uncommon disease through conducting a large, multi-center cohort study.

ELIGIBILITY:
Inclusion Criteria:

* within the age range of 18 to 65 years, diagnosed with rectal neuroendocrine tumors. Furthermore, patients were required to have a palpable tumor as determined by digital rectal examination or accessible through proctoscopy, with the distal border situated within 12 cm from the anal verge.

Exclusion Criteria:

* (1) muscularis propria invasion or NET grading = 3, (2)regional LN or distant organs metastasis at the time of diagnosis, (3) incomplete follow-up information, (4) the patient had multiple primary tumors, (5) patients with surgical excision or inappropriate methods such as forceps removal, and (6) the patient had a history of malignant tumors.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with rectal neuroendocrine tumors following initial endoscopic resection
Sampling Method: Probability Sample
Enrollment: 527 (Actual)
Dates: Start 2013-01-30 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
DFS | 5 year
  disease free survival

IPD SHARING:
Plan to Share IPD: No
available upon reasonable request